CLINICAL TRIAL: NCT03509285
Title: Randomized, Double-Blind, Double-Dummy, 5-Way Crossover Study to Evaluate the Abuse Potential of Cenobamate Relative to Alprazolam and Placebo When Administered Orally in Non-Dependent, Recreational Drug Users with Sedative Experience
Brief Title: A Study of the Abuse Liability Potential of Cenobamate in Recreational Drug Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: YKP3089C024
Record Dates: First submitted 2017-04-17; First posted 2018-04-26 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Alprazolam; Cenobamate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Qualification Y (Placebo Comparator): Placebo; administered orally as a single dose of 2 x 100 mg lactose tablets, over-encapsulated (alprazolam placebo)
  Interventions: Drug: Alprazolam Placebo
- Qualification Z (Active Comparator): Alprazolam 2.0 mg; administered orally as a single dose of 2 x 1.0 mg alprazolam tablets, over-encapsulated
  Interventions: Drug: Alprazolam
- Treatment A (Placebo Comparator): Placebo; administered orally as a single dose of 4 x cenobamate-matched placebo tablets and 3 x 100 mg lactose tablets, over-encapsulated (alprazolam placebo)
  Interventions: Drug: Alprazolam Placebo; Drug: Cenobamate placebo
- Treatment B (Active Comparator): Alprazolam 1.5 mg; administered orally as a single dose of 3 x 0.5 mg alprazolam tablets, over-encapsulated and 4 x cenobamate-matched placebo tablets
  Interventions: Drug: Cenobamate placebo; Drug: Alprazolam
- Treatment C (Active Comparator): Alprazolam 3.0 mg; administered orally as a single dose of 3 x 1.0 mg alprazolam tablets, over-encapsulated and 4 x cenobamate-matched placebo tablets
  Interventions: Drug: Cenobamate placebo; Drug: Alprazolam
- Treatment D (Experimental): Cenobamate, 200 mg; administered orally as a single dose of 2 x 100 mg cenobamate tablets, 2 x cenobamate-matched placebo tablets, and 3 x 100 mg lactose tablets, over-encapsulated (alprazolam placebo)
  Interventions: Drug: Alprazolam Placebo; Drug: Cenobamate placebo; Drug: Cenobamate
- Treatment E (Experimental): Cenobamate, 400 mg; administered orally as a single dose of 4 x 100 mg cenobamate tablets and 3 x 100 mg lactose tablets, over-encapsulated (alprazolam placebo)
  Interventions: Drug: Alprazolam Placebo; Drug: Cenobamate

INTERVENTIONS:
Drug: Alprazolam Placebo — 100 mg lactose tablets
  Arms: Qualification Y; Treatment A; Treatment D; Treatment E
Drug: Cenobamate placebo — Sugar pill manufactured to mimic cenobamate 100 mg tablet
  Arms: Treatment A; Treatment B; Treatment C; Treatment D
Drug: Alprazolam — 0.5 mg and 1.0 mg alprazolam tablets
  Arms: Qualification Z; Treatment B; Treatment C
Drug: Cenobamate — 100 mg tablet
  Arms: Treatment D; Treatment E

SUMMARY:
This randomized, single-dose, placebo- and active-controlled, crossover study will evaluate the abuse liability potential of cenobamate in recreational drug users with sedative drug use experience.

In the Qualification phase, subjects will receive a single dose of either alprazolam or placebo in a crossover design, with a wash-out period of at least 24 hours between treatments. Subjects who are clearly able to distinguish the positive control from placebo will be enrolled in the Treatment phase and will be randomized to single oral doses of cenobamate (2 dose levels), alprazolam (2 dose levels), and placebo in a double-blind, double-dummy, 5-way crossover design. Washout-periods between the 5 treatment periods in the Treatment phase will be at least 16 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects 18 to 55 years of age, inclusive.
2. Body mass index (BMI) within the range of 19.0 to 32.0 kg/m2, inclusive, and a minimum weight of 50.0 kg.
3. Current recreational drug users who have used benzodiazepines for recreational (non-therapeutic) purposes (i.e., for psychoactive effects) at least 5 times in the past year and used benzodiazepines at least once in the 12 weeks before Screening.
4. Female subjects of childbearing potential with male sexual partners must be using and willing to continue using medically acceptable contraception (as specified in Section 4.5.2) for at least 1 month prior to Screening (at least 3 months for oral and transdermal contraceptives) and for at least 30 days after the last study drug administration.
5. Female subjects of non-childbearing potential must meet the criteria specified in Section 4.5.2.
6. Male subjects with female sexual partners of childbearing potential must be using and willing to continue using medically acceptable contraception (as specified in Section 4.5.2) from Screening and for at least 30 days after the last study drug administration.
7. Able to speak, read, and understand English sufficiently to allow completion of all study assessments.
8. Must understand and provide written informed consent, prior to the initiation of any protocol-specific procedures.
9. Must be willing to comply with the requirements and restrictions of the study.

Exclusion Criteria:

1. Substance or alcohol dependence within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition - Text Revision (DSM IV-TR), and/or has ever participated or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence (excluding nicotine and caffeine).
2. Heavy smoker (>20 cigarettes per day) and/or is unable to abstain from smoking or unable to abstain from the use of prohibited nicotine-containing products for at least 10 hours during the in-clinic periods (including e-cigarettes, pipes, cigars, chewing tobacco, nicotine-topical patches, nicotine gum, or nicotine lozenges).
3. History or presence of clinically significant abnormality as assessed by physical examination, medical history (including cholecystectomy), ECGs, vital signs, or laboratory values, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results.
4. History or presence of myasthenia gravis, severe hepatic insufficiency, severe respiratory insufficiency, sleep apnea syndrome, or acute narrow angle glaucoma.
5. Positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
6. Evidence of clinically significant hepatic or renal impairment including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5× the upper limit of normal (ULN), or bilirubin >1× ULN. Repeat safety laboratory tests are allowed once for Screening, unless the principal investigator and sponsor agree to an additional repeat.
7. Donation or loss of more than 500 mL whole blood within 30 days preceding entry into the Treatment Phase.
8. Difficulty with venous access or unsuitable or unwilling to undergo catheter insertion.
9. Female subjects who are currently pregnant (have a positive pregnancy test) or lactating or who are planning to become pregnant within 30 days of last study drug administration.
10. History of severe allergic reaction (including anaphylaxis) to any substance, or previous status asthmaticus.
11. Subject history of allergy, hypersensitivity, or DRESS syndrome to any drug product including anti-convulsants (e.g., alprazolam, carbamazepine) or related drugs (e.g., other benzodiazepines) or known excipients of any of the drug products in this study. History of a first degree relative with a serious cutaneous drug-induced adverse reaction.
12. Subjects with any history of suicidal ideation or suicidal behavior, as assessed by the Columbia-Suicide Severity Rating Scale (C SSRS; baseline version).
13. Use of a prohibited medication or investigational drug, including exposure to any drugs associated with DRESS syndrome (e.g., allopurinol, minocycline, abacavir, lamotrigine) in the 6 months prior to Screening.
14. Use of a prohibited medication, as specified in Section 4.5.1.
15. Treatment with an investigational drug within 5 times the elimination half-life, if known (e.g., a marketed product), or within 30 days (if the elimination half-life is unknown) prior to the first study drug administration or is concurrently enrolled in any research judged not be scientifically or medically compatible with this study.
16. An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child or sibling, whether biological or legally adopted.
17. A subject who has pending legal charges or is on probation.
18. A subject who, in the opinion of the investigator or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason.
19. Anyone who has previously been exposed to cenobamate (prior to participation in this study).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-11-18 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics using Visual Analogue Scales (VAS) | Measured for 24 hrs in each Treatment Period
  Subjective Effect of Drug Liking "at this moment" [0-100 scale, 0=Strong Disliking, 50=Neither Like nor Dislike, 100=Strong Liking]

SECONDARY OUTCOMES:
Pharmacokinetics | Measured for 24 hrs in each Treatment Period
  Plasma concentrations of cenobamate and alprazolam
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 21 weeks
  Incidence, frequency, and severity of AEs and AEs of Special Interest (which include AEs related to drug reaction with eosinophilia and systemic symptoms [DRESS] and abuse-related adverse events)
Pharmacodynamics using Visual Analogue Scales (VAS) | Measured at 12 hr and 24 hr timepoints in each Treatment Period
  Subjective Effect of Take Drug Again [0-100 scale, 0=Definitely Not, 50=Neutral, 100=Definitely So]
Pharmacodynamics using Visual Analogue Scales (VAS) | Measured at 12 hr and 24 hr timepoints in each Treatment Period
  Subjective Effect of Overall Drug Liking [0-100 scale, 0=Strong Disliking, 50=Neither Like nor Dislike, 100=Strong Liking]
Pharmacodynamics using Visual Analogue Scales (VAS) | Measured for 24 hrs in each Treatment Period
  Subjective Effect of High [0-100 scale, 0=Not at All,100=Extremely]
Pharmacodynamics using Visual Analogue Scales (VAS) | Measured for 24 hrs in each Treatment Period
  Subjective Good Drug Effects [0-100 scale, 0=Not at All,100=Extremely]

CONTACTS AND LOCATIONS:
Locations (2):
- Vince & Associates Clinical Research, Inc, Overland Park, Kansas, United States
- INC Research, Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No